CLINICAL TRIAL: NCT06180863
Title: A Pilot Study of Oral Azacitidine (CC-486) Epigenetic Priming and Maintenance in Adult AML Patients Eligible for Reduced Intensity Allogeneic Stem Cell Transplant
Brief Title: Oral Azacitidine (CC-486) Epigenetic Priming and Maintenance for Adult Acute Myeloid Leukemia (AML) Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding.
Sponsor: Yale University (Other)
Collaborators: Bristol-Myers Squibb (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000031065; 1T32CA233414-01A1 (NIH)
Record Dates: First submitted 2023-11-17; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: Azacitidine; Reduced Intensity Allogeneic Stem Cell Transplant; Epigenetic priming; Complete remission
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Pathologic Complete Response | interventions — Azacitidine; cc-486

STUDY DESIGN:
Intervention Model Description: A single-arm non-randomized pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral azacitidine (CC-486) (Experimental): Patients on study will receive 300 mg CC-486 for 14 out of 28 days per cycle with dose modification according to the Onureg United States Prescribing Information (USPI). Up to 3 cycles of CC-486 will be allowed, and a minimum of 1 cycle is to be given prior to transplant. Multiple cycles will be allowed only if donor-specific or logistical issues prevent transplantation after the first cycle. CC-486 will be dispensed on day 1 of each treatment cycle and only 1 cycle equivalent is to be dispensed at the beginning of each cycle.
  Post-transplant maintenance with CC-486 can be started 60 days (range 60-120 days) after hematopoietic progenitor cell infusion which should allow time for count and graft recovery after post-transplant cyclophosphamide (PTCY). The CC-486 maximum preferred pre-emptive dose post-ASCT is 200 mg daily, which will be administered for 14 of 28 days per cycle (max 12 cycles).
  Interventions: Drug: oral azacitidine (CC-486)

INTERVENTIONS:
Drug: oral azacitidine (CC-486) — Oral azacitidine is indicated for continued treatment of adult patients with acute myeloid leukemia who achieved first complete remission (CR) or complete remission with incomplete blood count recovery (CRi) following intensive induction chemotherapy and are not able to complete intensive curative therapy.
  Other Names: Onureg

SUMMARY:
To investigate the feasibility of delivering oral azacitidine (CC-486) as a consolidation regimen from the time of first complete remission (CR1), in patients with acute myelogenous leukemia (AML) eligible for curative intent Allogeneic Stem Cell Transplant (ASCT).

DETAILED DESCRIPTION:
A significant proportion of patients with Acute myeloid leukemia (AML) who are fit to receive intensive chemotherapy and reach first complete remission (CR), relapse despite further high or low intensity therapies. Relapse/refractory (R/R) AML generally portends poor outcomes and available agents to treat this condition have modest efficacy. Until the recent approval of CC-486 as a maintenance therapy, no other drug had shown overall survival (OS) advantage for patients with AML in first complete remission (CR1). In the CC-486 registration trial (QUAZAR AML-01), remission induction was achieved by intensive chemotherapy, but patients were ineligible to proceed to allogeneic stem cell transplant (ASCT) at the time of screening. Post CR1, CC-486 apart from prolonging remission was also successful in deepening the quality of remission by eradicating measurable residual disease (MRD). It is therefore logical to investigate the feasibility of CC-486 as a consolidation regimen from the time of CR1, in patients eligible for curative intent ASCT. It is anticipated that continued epigenetic priming peri-ASCT with CC-486 can favorably alter disease biology for AML patients in CR1, modulate immune surveillance to decrease relapse risk, mitigate adverse graft versus host disease (GVHD) biology without significant compromise on the quality of life. This pilot study will assess the suitability of CC-486 as a bridge to transplant, will help optimize the timing between CC-486 administration and the start of transplant preparative regimen, and will assess the utility of continued CC-486 maintenance post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have acute myeloid leukemia (AML) of Intermediate or High risk (IR or HR per National Comprehensive Cancer [NCCN] Criteria) in first CR/CRi achieved with 1 or 2 cycles of cytarabine based induction therapy. Zero to 1 cycle of cytarabine based consolidation will be allowed post CR1. OR Nucleophosmin 1(NPM 1) positive AML ((in the absence of FMS like tyrosine kinase 3 (FLT3) mutation)) at diagnosis with positive NPM1 PCR (measurable residual disease [MRD]) after at least 1 cycle of cytarabine-based consolidation chemotherapy OR Secondary AML(s-AML) based on prior MDS or CMML in first CR/CRi. OR Therapy-related AML (t-AML) with IR or HR criteria
* Vyxeos induction (up to 2 cycles to reach CR1) and 0-1 cycle of vyxeos consolidation will be allowed.
* Eligible to receive RIC or Non myeloablative (NMA) transplant preparative regimen with post-transplant cyclophosphamide (PTCY) based GVHD prophylaxis, at the discretion of study investigator.
* Patients must have a calculated creatinine clearance (Cockcroft-Gault equation) > 50 mL/min.
* Patients must have a related or unrelated donor. Sibling donor must be a 6/6 match for human leukocyte antigen A (HLA-A) and HLA-B at intermediate or higher resolution, and DRB1 at high resolution using DNA-based typing; must be willing to donate peripheral blood stem cells; and meet institutional criteria for donation. Unrelated donor must be a 7/8 or 8/8 match at HLA-A, -B, -C, and -DRB1 at high resolution using DNA-based typing; must be willing to donate peripheral blood mononuclear cells (PBSCs); and be medically eligible to donate stem cells according to National Marrow Donor Program (NMDP) criteria.
* Patients must be willing to have peripheral blood stem cells as the graft source.
* Patients must have adequate hepatic function (i.e., serum bilirubin level ≤1.5 times the upper limit of normal [ULN], aspartate aminotransferase (AST), and alanine aminotransferase (ALT), defined as ≤2.5 × ULN). Higher levels of bilirubin are acceptable in the setting of Gilbert's disease with no other provable etiologies for altered liver function.
* Patients must have a Karnofsky performance score (KPS) ≥70 and/or ECOG score of ≤2.
* Patients must have recovered from the toxicities of the most recent induction/consolidation chemotherapy. Recovery is defined by the absence of persistent treatment-related AE of grade 2 or above. Persistent cytopenia meeting the criteria for a CRi and controlled infections on antimicrobials is acceptable.
* Women of childbearing potential must be surgically sterile or agree to practice abstinence or utilize acceptable contraception (intrauterine, injectable, transdermal, or combination oral contraceptive) during the period while receiving study medication and for at least 6 months after the last dose of CC-486. Males who are sexually active with women of childbearing potential must be surgically sterile or using an acceptable method of contraception (defined as barrier methods in conjunction with spermicides) from time of screening through at least 3 months after the last dose of CC-486.
* Patients must be able to understand the study procedures, agree to participate in the study program, and voluntarily provide written Informed Consent
* Patients must have no active COVID-19 infection symptoms at the time of enrollment. Those who tested positive in the past or made recovery post infection must be symptom free for at least 2 weeks prior to enrollment.
* Patients must be able to start transplant preparative regimens no later than 35 days from Day 1 of the most recent CC-486 cycle administration.

Exclusion Criteria:

* Patients may not have Acute Promyelocytic leukemia
* Patients may not have favorable risk AML per National Comprehensive Cancer Network (NCCN) guidelines ((Core binding factor leukemias, CCAAT/enhancer-binding protein-alpha (CEBPA) double mutant, AML with concomitant mutations in Nucleophosmin 1 (NPM1) and FLT3))
* Patients must not have received more than two rounds of chemotherapy to achieve first CR or CRi
* Patients may not have had exposure to hypomethylating agent (HMA) to treat the leukemia or prior hematologic malignancy ((i.e., myelodysplastic syndrome (MDS), Chronic Myelomonocytic Leukemia (CMML)) in the 6 months prior to study enrollment.
* Patients may not be, per investigator evaluation, currently in need of other leukemia-directed therapy such as FLT3- or Isocitrate dehydrogenase (IDH)-directed therapy.
* Patients may not have myeloproliferative neoplasm progressing to AML (except for CMML)
* With related and unrelated donors, patients may not have high pre-transplant donor-specific HLA antibodies warranting need for desensitization or other maneuvers per discretion of the treating physician.
* Patients may not have previously received radiation to maximum tolerable limits to any critical normal organ.
* Patients with prior Central Nervous System (CNS) involvement or extramedullary disease will be excluded.
* Patients may not have previously received allogeneic Hematopoietic Cell Transplantation (HCT).
* Patients may not have clinically significant cardiac disease ((New York Heart Association (NYHA) Class III or IV)); clinically significant arrhythmia i.e., ventricular tachycardia, ventricular fibrillation, or "Torsade de Pointes." Significant active cardiac disease within the previous 6 months including NYHA class 4 Congestive Heart Failure (CHF), Unstable angina, and Myocardial Infarction
* Patients may not have abnormal QTcF (>480 msec) after electrolytes have been corrected (at least two different ECG readings and at least 15 minutes between readings). Subjects with paced rhythm or prolonged QTcF may be exempt from this exclusion if considered eligible for transplant per treating physician clinical judgement with optional cardiology consultation.
* Patients may not have positive test results for human immunodeficiency virus (HIV) or hepatitis B (HBV) or C (HCV). Subjects with a past positive HBV test results due to previous exposure but who have cleared the virus or are vaccinated against hepatitis B, as evidenced by negative hepatitis B surface antigen (HbsAg), negative HBV viral load, and positive antibody to the HbsAg (anti-HBs) are not excluded. Subjects who have positive hepatitis test results with adequate organ function as defined in the protocol are not excluded.
* Patients may not have uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment)
* Patients may not have had an active malignancy within 1 year of entry. Active malignancy is defined as those malignancies requiring treatment with anti-cancer therapy or with a survival prognosis of less than 2 years at the time of inclusion. Exceptions to this exclusion include myelodysplastic syndrome/CMML, treated non-melanoma skin cancer, completely resected Stage 0 or 1 melanoma no less than 1 year from resection, cervical carcinoma in situ or cervical intraepithelial neoplasia, Breast cancers on long term hormonal therapy (1 year or more), and successfully treated organ-confined prostate cancer with no evidence of progressive disease based on prostate specific antigen (PSA) levels and not on active therapy.
* Patients may not be currently receiving any other investigational agents for relapse reduction.
* Patients seeking umbilical cord blood transplants, or bone marrow graft, or mismatched unrelated donor (MMUD) with <9/10 HLA match are ineligible.
* Ex-vivo T cell depletion or use of campath, antithymocyte globulin (ATG), or other anti-T cell antibodies as GVHD prophylaxis are not allowed. Patients are allowed to receive abatacept as approved by FDA.
* Patients may not have known uncontrolled and active alcohol or substance abuse
* Patients may not have any ongoing medical and non-medical condition that may render the patient ineligible for ASCT
* Pregnant or breast-feeding females are not eligible. (Lactating females must agree not to breast feed while taking CC-486).
* Patients may not have a history of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis), celiac disease (i.e., sprue), prior gastrectomy or upper bowel removal, or any other gastrointestinal disorder or defect that would interfere with the absorption, distribution, metabolism, or excretion of the study drug and/or predispose the subject to an increased risk of gastrointestinal toxicity
* Patients may not have abnormal coagulation parameters (PT >15 seconds, PTT>40 seconds, and/or INR >1.5). Patients with chronic anticoagulation can be considered for inclusion after discussion with the PI
* Patients may not have known or suspected hypersensitivity to azacitidine or mannitol
* Patients may not have any significant medical, surgical, or mental health problem that would prevent appropriate patient participation in the study
* Patients may not have any conditions including, but not limited to, laboratory abnormalities which put patients at unacceptable risk as per evaluation of treating physician
* Patients may not have a history of idiopathic thrombocytopenic purpura, disseminated intravascular coagulation, thrombotic thrombocytopenic purpura (TTP) or hemolytic uremic syndrome (HUS)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients receiving oral azacitidine (CC 486) as post-remission consolidation therapy that are able to proceed to reduced intensity conditioning (RIC) allogeneic stem cell transplant (ASCT) | With each cycle (1 cycle is equivalent to 28 days) of CC-486 pre-transplant, up to 3 months
  To identify the number of participants able to receive a minimum of 1 and a maximum of 3 cycles of CC-486 consolidation therapy as a bridge to Reduced Intensity Conditioning (RIC) ASCT while maintaining first complete remission- CR1.
Total number of participants that experience any adverse events with oral azacitidine (CC 486) use prior to RIC ASCT for patients with (AML) in first complete remission (CR1). | For a maximum of 3 cycles (1 cycle is equivalent to 28 days) and or up to 3 months from the start of CC-486
  Adverse events (AEs) occurring in the participants will be graded according to NCI CTCAE v 5.0 with each cycle of CC_486 administered pre-transplant.

SECONDARY OUTCOMES:
Disease status and response to each cycle of pre-transplant CC-486 administration as per European Leukemia Net (ELN) AML 2017 guidelines | With each cycle (1 cycle is equivalent to 28 days) of CC-486 pre-transplant
  With CC-486 consolidation prior to transplant best response to treatment and disease status will be measured. Response criteria or loss of response (including frank morphologic relapse) will be assessed by using peripheral blood or bone marrow samples as per European Leukemia Net (ELN) AML 2017 guidelines.
Number of participants retaining remission post-transplant | Up to 720 days
  Bone marrow biopsies will be performed longitudinally post-transplant. Prior to initiating first cycle of CC-486 maintenance post-transplant, disease status confirmation with a bone marrow biopsy in the prior 14 days would be needed. Response criteria or loss of response will be defined as per European Leukemia Net (ELN) AML 2017 guideline. Based on best response observed duration of remission, cumulative incidence of relapse, patterns of relapse will be described. Participants will be assessed at days 30, 60, 120, 180, 365 and 720 for disease relapse.
Total number of maintenance cycles administered post-transplant to assess compliance | Up to 2 years post transplant
  As assessed by the number of cycles administered and the periods of interruptions.
Overall Survival | Up to 2 years from the time of starting CC-486
  As assessed by the length of survival in months from the time of 1st cycle of CC-486 pretransplant, from the time of transplant and from the time of starting maintenance post-transplant.
Incidence of graft versus host disease (GVHD) | up to 2 years post-transplant
  As assessed by cumulative incidence of acute and chronic graft versus host disease (GVHD) within 2 years from the date of transplant.
Hematopoiesis origins assessed in peripheral blood and bone marrow. | Up to 2 years post transplant
  As assessed by kinetics of chimerism changes for those receiving CC-486. Based on institutional practices peripheral blood and or bone marrow samples would be used for chimerism testing. Donor/recipient hematopoiesis fraction will be reported across cellular subset per institutional standards.
Change in quality of life assessed by Foundation for the Accreditation of Cellular Therapy Bone Marrow Transplant (FACT-BMT) version 4. | Prior to transplant (at screening and immediately prior to transplant) and in post-transplant at days + 100, +180 & +365
  Quality of life questionnaire administered pre- and post-transplant with CC-486 maintenance use. The Likert scale from zero to four [0-4] is used to measure the responses for each question after taking into account reverse scores for questions constructed in a negative form. The final score for FACT-BMT ranges from zero to 196. Higher scores for the scales and subscales indicate better quality of life.
Total number of participants that experience any adverse events with oral azacitidine (CC 486) use in post-transplant period. | up to 2 years post transplant
  Adverse events (AEs) occurring in the participants will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v 5.0 with each cycle of CC_486 administered post-transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Lohith Gowda, MD, Principal Investigator — Yale University; Marcos de Lima, MD, Principal Investigator — Ohio State University
Locations (1):
- Yale Comprehensive Cancer Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No